CLINICAL TRIAL: NCT01503775
Title: A Prospective, Multicentric Observational Study Evaluating the Long Term Efficacy and Safety of the CODMAN TRUFILL®'s Line of Coils in the Endovascular Treatment of Intracranial Aneurysms
Brief Title: TRUfill®'s Line in Intracranial aNeurysm Embolisation
Acronym: TRULINE
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-PMK-0902
Record Dates: First submitted 2011-12-23; First posted 2012-01-04 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Aneurysms
Keywords: intracranial; ruptured; non-ruptured; aneurysms; Intracranial ruptured or non-ruptured aneurysms
MeSH Terms: conditions — Aneurysm; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TRUFILL® DCS Orbit Galaxy

SUMMARY:
The objective of this study is to evaluate the long term efficacy and safety of the CODMAN TRUFILL®'s line of coils in the treatment of patients with intracranial ruptured or non-ruptured aneurysms in real-life routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient presenting one or more ruptured or non-ruptured intracranial aneurysms assessed by angiography
* Patient implanted with one or more CODMAN TRUFILL® coils
* Patient agree to take part in the study, or agreement of a representative of the patient in case of patient inability, after being informed by the investigator and have received information letter.

Exclusion Criteria:

* Patient who does not accept to take part in the study after being informed
* Patient already enrolled in a clinical trial involving experimental medication or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
The long term safety of the coiling procedure with the CODMAN TRUFILL®'s line of coils will be assessed by the combined morbidity-mortality rate (CMMR) observed during the procedure and up to 1 year post-procedure follow-up. | Observed during the procedure and up to 1 year post-procedure follow-up

SECONDARY OUTCOMES:
The procedural CMMR observed during the procedure and up to 30 Days post procedure follow-up. | Observed during the procedure and up to 30 Days post procedure follow-up.
The rate of permanent morbidity and mortality observed at 30 Days and at 1 year post-procedure follow-up, defined as a mRS of 3 to 6. | Observed at 30 Days and at 1 year post-procedure follow-up
The rate of absence of deterioration or improvement of the neurological status observed at 30 days and at 1 year post procedure follow-up | Observed at 30 days and at 1 year post procedure follow-up
The overall rate of Adverse Event/Serious Adverse Event observed during the procedure, at 30 days and up to 1 year post-procedure follow-up | Observed during the procedure, at 30 days and up to 1 year post-procedure follow-up
The rate of Adverse Event/Serious Adverse Event related to the device and/or to the procedure observed during the procedure, at 30 days and up to 1 year post-procedure follow-up | Observed during the procedure, at 30 days and up to 1 year post-procedure follow-up
The rate of Unanticipated Adverse Device Effects observed during the procedure, at 30 days and up to 1 year post-procedure follow-up | Observed during the procedure, at 30 days and up to 1 year post-procedure follow-up
The rate of per-procedural subarachnoid hemorrhage of the treated aneurysm and rate of per-procedural SAH leading to a modification of the procedure initially planned | During the procedure
The rate of recurrent subarachnoid hemorrhage of the treated aneurysm at one-year post-procedure follow-up | 1 year post-procedure
The rate of aneurysm occlusion at the end of the procedure and at 1 year post-procedure follow-up | End of the procedure and at 1 year post-procedure follow-up
The rate of aneurysm recanalisation up to 1 year post-treatment defined as any increase in the size of the remnant or defined as a change of classification of the Raymond scale result related up to the 1 year post-procedure follow-up | Up to 1 year post-treatment
The rate of spontaneous aneurysm regression up to 1 year post-treatment defined as any decrease in the size of the remnant or defined as a change of classification of the Raymond scale result related up to the 1 year post-procedure follow-up | Up to the 1 year post-procedure follow-up
The rate of retreatment at 1 year follow-up representing the rate of major recurrence on the target aneurysm observed up to the 1 year post-procedure follow-up | Up to the 1 year post-procedure follow-up

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Hôpital Neurologique, Lyon
  - Clinique Clairval, Marseille
  - Hôpital Adullte La Timone, Marseille
  - Fondation Rothschild, Paris
  - CHU Pontchaillou, Rennes